CLINICAL TRIAL: NCT01798810
Title: Supplemental Perioperative Oxygen to Reduce Surgical Site Infection After High Energy Fracture Surgery (OXYGEN Study)
Brief Title: Supplemental Perioperative Oxygen to Reduce Surgical Site Infection After High Energy Fracture Surgery
Acronym: OXYGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-12-1-0588
Record Dates: First submitted 2013-02-18; First posted 2013-02-26 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Surgical Site Infection
Keywords: Surgical Site Infection Risk Prediction; Bacterial species type and antibacterial sensitivities; Resource Utilization and Cost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental Perioperative Oxygen (80% FiO2) (Experimental): After intubation, patients in the Treatment Group will receive intraoperative inspired oxygen set at 80 percent (FiO2 of 0.80). Post-extubation, patients in the treatment arm will be placed on high flow non-re-breather mask at 15L/min for up to 2 hours postoperatively and then transitioned to nasal cannula, which will be weaned as tolerated.
  Interventions: Procedure: Supplemental Perioperative Oxygen
- Control (30% FiO2) (No Intervention): After intubation, patients in the control arm will receive typical standard of care intraoperative inspired oxygen of 30 percent (FiO2 of 0.30). Post-extubation, patients in the control arm of the study will be placed on a nasal cannula at 4L/min to maintain SaO2≥92% as determined by pulse oximetry. This will be maintained for up to 2 hours and then weaned as tolerated.

INTERVENTIONS:
Procedure: Supplemental Perioperative Oxygen — Patients receiving perioperative oxygen will receive 80% FiO2 during surgery.
  Arms: Supplemental Perioperative Oxygen (80% FiO2)

SUMMARY:
The OXYGEN Study is a double blinded prospective randomized controlled trial that will compare the proportion of surgical site infections within 6 months in patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

DETAILED DESCRIPTION:
Primary Objective

To compare the proportion of surgical site infections within 6 months in patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

Secondary Objectives

To compare species and antibacterial sensitivities of the bacteria in the patients who develop surgical site infections in study patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

To validate the previously developed risk prediction model for the development of surgical site infections after fracture surgery

To measure and compare resource utilization and cost associated with surgical site infection in study patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

Primary Aim: To compare the proportion of surgical site infections within 6 months in patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

Hypothesis 1: The proportion of surgical site infections will be lower for patients treated with Supplemental Perioperative Oxygen.

Secondary Aim #1: Compare bacterial species and antimicrobial susceptibilities in the patients who develop surgical site infections in study patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

Hypothesis 2: In the patients who develop infections, the bacterial species and antimicrobial susceptibility profiles of those treated with Supplemental Perioperative Oxygen will be similar to those treated without Supplemental Perioperative Oxygen.

Secondary Aim #2: To validate the previously developed risk prediction model for the development of surgical site infections after fracture surgery.

Hypothesis 3: The previously developed RIOTS score will be highly predictive of infection risk.

Secondary Aim #3: Measure and compare resource utilization and cost associated with surgical site infection in study patients treated with Supplemental Perioperative Oxygen compared to those treated without Supplemental Perioperative Oxygen.

Hypothesis 4: Supplemental Perioperative Oxygen will be associated with lower resource utilization and cost.

ELIGIBILITY:
Inclusion Criteria:

* All "high energy" tibial plateau fractures treated operatively with plate and screw fixation. We define "high energy" tibial plateau fractures as patients who are either:

  * Initially treated with an external fixation and treated more than 7 days later after swelling has resolved.
  * Gustilo Type I, II, and IIIA open fracture, regardless of timing of definitive treatment.
* All "high energy" pilon (distal tibial plafond) fractures treated operatively with plate and screw fixation. We define "high energy" tibial plateau fractures as patients who are either:

  * Initially treated with an external fixation (with or without fibula fixation or limited internal fixation) and treated definitively more than 7 days later after swelling has resolved.
  * Gustilo Type I, II, and IIIA open fracture, regardless of timing of definitive treatment.
* All "high energy" calcaneus fractures treated operatively with plate and screw fixation in a staged fashion. We define "high energy" calcaneus fractures as patients who are either:

  * Treated definitively more than 7 days later after swelling has resolved.
  * Gustilo Type Type I, II, and IIIA [30,31] open fracture, regardless of timing of definitive treatment.
* Ages 18 to 80 years
* Patients may have co-existing infection not at study fracture site, with or without antibiotic treatment.
* Patients may have risk factors for infection including diabetes, immunosuppression from steroids or other medications, HIV, or other infections.
* Patients may have a head injury.
* Patients may be treated initially with a temporary external fixator prior to randomization.
* Patients may have a portion of the fixation (e.g. fibula fixation in pilon or percutaneous screws across a tibial plateau fracture) prior to definitive plate fixation, at any initial surgery before randomization for definitive fixation.
* Patients may have other orthopedic and non-orthopaedic injuries.
* Patients may have pre-existing musculoskeletal injuries, be non ambulators, or have spinal cord injuries.

Exclusion Criteria:

* Tibial plateau, pilon, or calcaneus already infected at time of study enrollment.
* Type IIIB, or IIIC open [30,31] fractures
* Patient speaks neither English nor Spanish.
* Transfer patients who have already had definitive fixation.
* Severe problems with maintaining follow-up (e.g. patients who are homeless at the time of injury or those how are intellectually challenged without adequate family support).
* Patients who are intubated at the time of consent.
* Patients whose oxygen requirements at the time of surgery would prevent them from participating in either study group will be excluded.
* History of COPD or any other chronic respiratory disease that renders the patient oxygen dependent at baseline.
* Current or history of Bleomycin use (chemotherapy use associated with oxygen toxicity).
* Patient is currently pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-06; Primary Completion 2019-05 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection | 26 weeks
  The main outcome measure will be the presence of clinically significant surgical site infection (SSI) in the first 26 weeks after surgery, as determined by CDC guidelines.
  Wound characteristics will also be evaluated using the ASEPSIS score. In this system wounds are scored using the weighted sum of points assigned for predetermined criteria including the need for Additional treatment, presence of Serous drainage, Erythema, Purulent exudates, Separation of deep tissues, the Isolation of bacteria, and the duration of patients Stay (ASEPSIS).

SECONDARY OUTCOMES:
Catalog and Compare Bacterial Species | 26 weeks
  Secondary outcome measures in this study include culture data in the group that becomes infected. Sensitivities of the isolated bacteria, which are also determined routinely in current clinical practice, will be recorded for analysis.
  We will also describe the type of antibiotic resistance experienced in both groups. There are 3 specific types of antibiotic resistance that will be analyzed. These have been chosen because they are currently of most clinical importance in the treatment of surgical site infection after civilian fracture surgery.
  * MRSA: Methicillin resistance staph aureus rates will be analyzed.
  * VRE: Vancomycin resistant enterococcus rates will be analyzed.
  * MDR GNR: Multi drug resistant gram negative rates will be analyzed.
Risk Factors for Infection | 26 weeks
  Our previous work in the pilot study allowed us to propose a novel score to the risk of surgical site infection after high energy fracture surgery: the RIOTS (Risk of Infection for Orthopaedic Trauma Surgery. We will attempt to better validate our previous score on this larger multi-center dataset and further investigate if other risk factors for infection should be included.
  Data collected includes all demographic characteristics of the patient, the descriptors of the injury, and details of the surgical treatment that would be available prior to the definitive surgery will be collected for analysis regarding determination of a model to predict infection risk in this patient population. These factors have been defined in previous work by this study team.
Resource Utilization and Cost | 1 year
  Previous research has shown that SSI increases length of stay and overall cost of treatment for surgery patients. Three data sets in the case report forms will be used to document medical resource utilization associated with surgical site infections in this trial: initial hospital admission, hospital readmission for SSI, and follow-up visit forms. During scheduled follow-up visits study participants will be queried regarding post-discharge treatment that may be associated with SSI such as antibiotic infusion therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Renan Castillo, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health; Robert O'Toole, MD, Principal Investigator — University of Maryland R Adams Cowley Shock Trauma Center; Anthony Carlini, MS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Banner University Medical Center/The CORE Institute, Phoenix, Arizona
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland